CLINICAL TRIAL: NCT05904496
Title: A Phase 1a/1b Study Investigating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of the DGKζ Inhibitor BGB-30813, Alone or in Combination With the Anti-PD-1 Monoclonal Antibody Tislelizumab in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study of BGB-30813 Alone or in Combination With Tislelizumab in Participants With Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor has made the decision to discontinue the clinical development of BGB-30813 and close the study based on imbalanced benefit/risk profile in the BGB-A317-30813-101 study.
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-30813-101; U1111-1290-6118 (Other: WHO); 2023-503996-38 (EudraCT Number); CTR20233404 (Other: ChinaDrugTrials)
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors
Keywords: DGKζ Inhibitor; BGB-30813; Anti-PD-1 Monoclonal Antibody; Tislelizumab; Advanced or Metastatic Solid Tumors; Diacylglycerol kinase; BGB-A317; NSCLC; Immunotherapy; HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1a: Dose Escalation Part A: BGB-30813 Monotherapy (Experimental)
  Interventions: Drug: BGB-30813
- Phase 1a: Dose Escalation Part B: BGB-30813 + Tislelizumab (Experimental)
  Interventions: Drug: BGB-30813; Drug: Tislelizumab
- Phase 1b: Dose Expansion BGB-30813 in Combination with Tislelizumab (Experimental)
  Interventions: Drug: BGB-30813; Drug: Tislelizumab

INTERVENTIONS:
Drug: BGB-30813 — Specified dose administered on specified days
Drug: Tislelizumab — Specified dose administered on specified days
  Other Names: BGB-A317
  Arms: Phase 1a: Dose Escalation Part B: BGB-30813 + Tislelizumab; Phase 1b: Dose Expansion BGB-30813 in Combination with Tislelizumab

SUMMARY:
This is a First in Human (FIH) Phase 1, multicenter, open label, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary antitumor activity of BGB-30813 as monotherapy or in combination with tislelizumab in participants with advanced or metastatic solid tumors. The study will be conducted in 2 parts: Phase 1a dose escalation and Phase 1b dose expansion.

DETAILED DESCRIPTION:
This study will test whether taking BGB-30813 alone or with tislelizumab can help treat patients with cancer that has spread throughout the body or is locally advanced. The two main goals of the study are to ensure that the treatments are safe by monitoring side effects and to determine the number of participants who respond well to treatment either partially or completely. The combination of BGB-30813 with other drugs that target immune checkpoints may work together to stop or prevent cancer activity.

Approximately 200 participants will participate. In the first part of the study, participants will be given different doses of BGB-30813 either alone or with tislelizumab to find the dose that is best tolerated. BGB-30813 will be given orally and tislelizumab will be given through a vein. In the second part of the study, the selected dose of BGB-30813, either alone or with tislelizumab, will be given to a larger number of participants from different parts of the world to see if the treatments can improve the signs and symptoms of their cancer. Treatments will continue until participants are no longer considered to be receiving benefits, have unacceptable side effects, or withdraw consent.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1a (Dose Escalation):

  * Participants with histologically or cytologically confirmed advanced, metastatic, and unresectable solid tumors who have previously received available standard systemic therapy or for whom treatment is not available or not tolerated and who have not received any prior therapy targeting diacylglycerol kinase (DGK)
  * Eligible tumor types are immune sensitive solid tumors such as non-small cell lung cancer (NSCLC), head neck squamous cell cancer (HNSCC), small cell lung cancer, hepatocellular carcinoma, esophageal cancer, gastric or gastroesophageal carcinoma, nasopharyngeal carcinoma, triple-negative breast cancer, urothelial carcinoma, renal cell carcinoma, cervical cancer, endometrial carcinoma, cutaneous squamous cell carcinoma, melanoma, Merkel cell carcinoma, mesothelioma, microsatellite instability (MSI)-high, tumor mutation burden (TMB)-high, or mismatch repair deficient solid tumors
  * Prior checkpoint inhibitor (CPI) therapy is allowed
* Phase 1b (Dose Expansion):

  * Participants with selected advanced or metastatic solid tumors including NSCLC, HNSCC, and additional potential tumor types to be defined based on emerging data
* ≥ 1 measurable lesion per RECIST v1.1
* Eastern Cooperative Group Oncology Performance (ECOG) Performance Status score ≤ 1
* Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study
* Adequate organ function as indicated by the following laboratory values up to first dose of study treatment: Hemoglobin≥ 90 grams per liter (g/L), Absolute neutrophil count ≥ 1.5 x 109/L , Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) (< 3 x ULN for participants with Gilbert syndrome ), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN

Exclusion Criteria:

* Previous therapy targeting DGK
* Active leptomeningeal disease or uncontrolled symptomatic central nervous system (CNS) metastasis
* Active autoimmune diseases or history of autoimmune diseases that may relapse
* Any active malignancy ≤ 2 years before the first dose of study treatment except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent
* Systemic anticancer therapy, including chemotherapy ≤ 21 days or 5 half-lives (whichever is shorter) before the first dose of study drugs
* ≥ Grade 3 immune-mediated adverse events on prior immuno-oncology agent (anti-PD-1 or anti-CTLA4 antibodies or other experimental drugs)

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Phase 1a: Dose Escalation: Number of Participants Experiencing Adverse Events (AEs), Serious Adverse Events (SAEs) and Dose-Limiting Toxicities (DLTs) | From the first dose of study drug(s) to 30 days after the last dose; approximately 6 months
  Number of participants experiencing AEs and SAEs, including physical examination findings, electrocardiograms (ECGs), and lab assessments as needed; and AEs meeting protocol-defined DLT criteria.
Phase 1a: Dose Escalation: The Maximum Tolerated Dose (MTD) and Maximum Administered Dose (MAD) | Up to approximately 6 months
  The MTD or MAD is defined as the highest dose at which 30% of participants experience a DLT or the highest dose administered, respectively.
Phase 1a and 1b: Recommended dose(s) for Expansion (RDFE[s]) of BGB-30813 Alone or in Combination with Tislelizumab | Up to approximately 6 months
  The RDFE(s) of BGB-30813 alone or in combination with tislelizumab, determined based upon the MTD or MAD and other relevant data.
Phase 1b: Dose Expansion: Overall Response Rate (ORR) as Determined by the Investigator | Up to approximately 12 months
  ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) as determined from tumor assessments by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Phase 1a: Dose Escalation: ORR as Determined by the Investigator | Up to approximately 12 months
  ORR is defined as the percentage of participants who had confirmed CR or PR as determined from tumor assessments by the investigator per RECIST version 1.1
Phase 1a: Dose Escalation: Maximum Observed Plasma Concentration (Cmax) Of BGB-30813 and Metabolite BGB-33481 Alone and in Combination with Tislelizumab | Up to approximately 6 months
Phase 1a: Dose Escalation: Observed Plasma Trough Concentration (Ctrough) Of BGB-30813 and Metabolite BGB-33481 Alone and in Combination with Tislelizumab | Up to approximately 6 months
Phase 1a: Dose Escalation: Area under the concentration-time curve (AUC) Of BGB-30813 and Metabolite BGB-33481 Alone and in Combination with Tislelizumab | Up to approximately 6 months
Phase 1a: Dose Escalation: Half-life (t1/2) Of BGB-30813 and Metabolite BGB-33481 Alone and in Combination with Tislelizumab | Up to approximately 6 months
Phase 1b: Dose Expansion: Number of Participants Experiencing AEs and SAEs | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 6 months
  Number of participants experiencing AEs and SAEs, including physical examination findings, ECGs, and lab assessments as needed.
Phase 1b: Dose Expansion: Duration of Response (DOR) | Up to approximately 12 months
  DOR is defined as the time from the first determination of an overall response assessed by the investigator using RECIST v1.1, until the first documentation of disease progression or death, whichever comes first.
Phase 1b: Dose Expansion: Disease Control Rate (DCR) | Up to approximately 12 months
  DCR is defined as the percentage of participants with best overall response (BOR) of complete Response (CR), Partial Response (PR), or stable disease assessed by the investigator using RECIST v1.1.
Phase 1b: Dose Expansion: Progression Free Survival (PFS) | Up to approximately 12 months
  PFS is defined as the time from the date of the first dose of study drugs to the date of the first documentation of disease progression assessed by the investigator using RECIST v1.1 or death, whichever occurs first.
Phase 1b: Dose Expansion: Clinical Benefit Rate (CBR) | Up to approximately 12 months
  CBR is defined as the percentage of participants with BOR of confirmed CR, PR, or stable disease lasting ≥ 24 weeks as assessed by the investigator using RECIST v1.1.
Phase 1b: Dose Expansion: Plasma concentrations of BGB-30813, and its metabolite, BGB-33481 | Up to approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (11):
- United States (3):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Md Anderson Cancer Center, Houston, Texas
  - Next Oncology, San Antonio, Texas
- Australia (3):
  - Monash Health, Clayton, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- China (3):
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
- Spain (2):
  - Hospital Universitario Vall Dhebron, Barcelona
  - Start Madrid Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/